CLINICAL TRIAL: NCT02899065
Title: Evaluation of the Roche Cobas Liat Flu/RSV Assay for Management of Influenza in the Emergency Department
Brief Title: Evaluation of the Roche Liat Flu/RSV Assay for Management of Influenza in the Emergency Department
Acronym: Influenza
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 906232
Record Dates: First submitted 2016-08-02; First posted 2016-09-14 (Estimated); Results first posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention (Experimental): The intervention arm will receive pharmacist-led education and stewardship intervention and a procalcitonin test to aid in the decision of how to treat the patient. This intervention will include direct delivery of education from the pharmacist to the treating clinician about interpreting the Roche Cobas Liat Flu/RSV and procalcitonin test results, recommendations for antiviral-treatment for high-risk patients and information about infection control precautions for patients being hospitalized with a positive RSV or influenza test.
  Interventions: Diagnostic Test: Procalcitonin; Other: Pharmacist-Led Education
- Standard of care (No Intervention): The second arm will be usual care (i.e. Roche Cobas Liat Flu/RSV test only). Results will be delivered via standard of care.

INTERVENTIONS:
Diagnostic Test: Procalcitonin — Procalcitonin is a blood test used to differentiate between viral and bacterial infections. This test is expected to aid in determining the best course of treatment for patients enrolled into this arm.
  Arms: Intervention
Other: Pharmacist-Led Education — Pharmacists will interpret the results of the Roche Cobas Liat Flu/RSV assay and procalcitonin test (if available) and provide the treating physician with recommendations for antibiotic therapy based on these results.
  Arms: Intervention

SUMMARY:
This will be a prospective, patient-oriented, pilot randomized clinical trial to evaluate (in aggregate) both the use of the Roche Cobas Liat Flu/RSV Assay and the use of pharmacist-led education for providers in the interpretation of these test results.

DETAILED DESCRIPTION:
To determine if pharmacist-led education and procalcitonin testing as part of a stewardship intervention optimizes antiviral treatment and reduces antibiotic treatment for pediatric Emergency Department (ED) patients with suspected influenza v. standard care (i.e. rapid molecular influenza test without patient specific treatment recommendations) using a prospective, patient-randomized design.

Consented patients in the pediatric ED will be randomized into two arms: The intervention arm will receive a patient specific stewardship intervention and procalcitonin testing during the ED visit. The intervention will be pharmacist-led and include direct delivery to clinicians of information about interpreting test results and recommendations for antiviral-treatment for high-risk patients, and infection control precautions for patients being hospitalized with a positive RSV or influenza test. Clinician adherence to treatment guidelines with and without the educational intervention will be compared.

The second arm will be usual care (i.e. no procalcitonin test or pharmacist-led education). Results will be delivered via standard of care through the electronic medical record (EMR).

Physicians and patients will not be blinded to arm assignments. Tests will be performed on a real-time basis in the ED. For each of these groups, data of the frequency and duration of antibiotic administration, antiviral use, adherence to evidence based guidelines for treatment of influenza, isolation, hospitalizations, and unscheduled return visits or readmissions within a 30 day period will be collected and compared.

Research coordinators will contact patients and/or parents at 1 and 4 weeks after enrollment for self-reported secondary outcomes including symptom resolution, return to school/work, and follow up healthcare visits, medication adherence (to antibiotics and/or antivirals), and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients <50 years of age who are evaluated in the emergency department for:
* suspected influenza, including symptoms of influenza-like illness (ILI - including fever > 38 degrees Celsius and cough or sore throat), or
* non-specific upper respiratory infection (URI) for whom the clinician suspects the presence of RSV, or influenza, or lower respiratory infection LRI).
* Patients whose treating provider has ordered a Roche Cobas Liat Flu/RSV test.

Exclusion Criteria:

* Patients who are pregnant
* Prisoners
* Patients who are unable to give informed consent in English or Spanish.
* Provider is unwilling to wait for procalcitonin results.

Max Age: 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larissa S May, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/evaluation-of-a-medical-test-for-management-of-the-flu-in-the-emergency-department-400713/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited after presentation to the Emergency Department between March 2018 and April 2022 at the University of California Davis Medical Center.
Pre-assignment Details: During the enrollment period, 1259 ED patients were assessed for inclusion and 200 were randomized into the research study.
Groups:
- Intervention Arm: Participants enrolled to the intervention arm received a procalcitonin lab test along with the standard of care Roche Cobas Liat Flu/RSV lab testing. The intervention also included pharmacist-led education and stewardship to the treating clinician about interpreting the Roche Cobas Liat Flu/RSV and procalcitonin test results, recommendations for antiviral-treatment for high-risk patients, and information about infection control precautions for patients being hospitalized with a positive RSV or influenza test.
- Standard of Care: This arm consisted of the delivery of Emergency Department usual care (i.e. Roche Cobas Liat Flu/RSV test only). Results were delivered via standard of care reporting.
Period: Randomization to 7 Day Follow Up Contact
Arm/Group | Intervention Arm | Standard of Care
Started | 100 (Procalcitonin results available: n=93 Procalcitonin results not available: n=7) | 100 (Procalcitonin results available: n=33 Procalcitonin results not available: n=67)
Completed | 99 | 95
Not Completed | 1 | 5
Not completed — Withdrawal by Subject | 1 | 5
Period: Day 7 to 4 Week Follow Up Contact
Arm/Group | Intervention Arm | Standard of Care
Started | 99 | 95
Completed | 75 | 79
Not Completed | 24 | 16
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lost to Follow-up | 21 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Standard of Care | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: months] | 149 (157) | 124 (140) | 136 (149)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 47 | 91
  Male | 56 | 53 | 109
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 49 | 46 | 95
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 200
Education - n = Some college [Count of Participants; unit: Participants] | 16 | 11 | 27
Height [Mean (Standard Deviation); unit: inches] — Population: Not all patients who present to the ED have their height measured; therefore, a portion of the study population do not have a recorded height.
  inches
    number analyzed (Participants) | 80 | 77 | 157
    (all) | 50.5 (16.5) | 50.8 (14.9) | 50.7 (15.7)
Weight [Mean (Standard Deviation); unit: kilograms] — Population: Not all patients who present to the ED are weighed; therefore, a small portion of the study population do not have a recorded weight.
  kilograms
    number analyzed (Participants) | 99 | 97 | 196
    (all) | 40.0 (33.7) | 38.7 (34.6) | 39.3 (34.1)
Temperature [Mean (Standard Deviation); unit: celsius] — Population: One participant did not have a recorded temperature.
  celsius
    number analyzed (Participants) | 100 | 99 | 199
    (all) | 37.7 (1.1) | 37.6 (1.0) | 37.6 (1.0)
Influenza A positive [Count of Participants; unit: Participants] | 13 | 11 | 24
Influenza B positive [Count of Participants; unit: Participants] | 8 | 5 | 13
Respiratory syncytial virus - RSV positive [Count of Participants; unit: Participants] | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Prescribed Antibiotics
Description: The determination of whether use of the Roche Cobas/Liat Flu/RSV Assay as part of a stewardship intervention reduces antibiotic treatment for pediatric ED patients with suspected influenza. Proper adherence to treatment guidelines after results should reduce physician prescription of antibiotic for non-responsive conditions.
Time Frame: During ED stay, up to 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Standard of Care
Number analyzed (Participants) | 100 | 100
Participants | 39 | 32

2. Primary Outcome: Number of Participants Prescribed Antiviral Therapy
Description: The determination of whether use of the Roche Cobas Liat Flu/RSV Assay as part of a formal stewardship intervention optimizes antiviral treatment of pediatric ED patients with influenza at risk of complications.
Time Frame: During ED stay, up to 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Standard of Care
Number analyzed (Participants) | 100 | 100
Participants | 12 | 10

3. Secondary Outcome: Emergency Department Recidivism
Description: Emergency Department return visits within 30 days for patients diagnosed with influenza and RSV
Time Frame: 30 days
Population: Number of participants who tested positive during their initial ED visit
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Standard of Care
Number analyzed (Participants) | 28 | 23
Participants | 19 | 16

4. Secondary Outcome: Symptom Resolution
Description: Time to resolution of symptoms such as fever, cough or sore throat
Time Frame: 7 days and again at week 4
Population: The total participants randomized in the study was 200 with an equal number in both arms (100). Of the 100 participants randomized to each arm, only 87 were able to be contacted in the intervention arm and 82 participants in the standard of care arm at Day 7. At week 4, 76 participants were able to be contacted in the intervention arm and 77 were contacted in the standard of care arm. The remaining participants were either lost to follow up or withdrew consent for participation in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Standard of Care
Number analyzed (Participants) | 87 | 82
Participants
  Symptoms Resolved by Day 7 | 66 | 52
  Symptoms resolved by Week 4: number analyzed (Participants) | 76 | 77
  Symptoms resolved by Week 4 | 62 | 61

5. Secondary Outcome: Lost Days of School/Work
Description: Number of days of school and/or work missed due to illness
Time Frame: 7 days and again at week 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Intervention Arm | Standard of Care
Number analyzed (Participants) | 87 | 82
Days
  School days missed at day 7 | 2.6 (3.0) | 2.6 (3.1)
  Work days missed at day 7 | 2.5 (2.7) | 3.1 (3.1)
  School days missed at week 4: number analyzed (Participants) | 76 | 77
  School days missed at week 4 | 1.8 (3.7) | 1.4 (4.1)
  Work days missed at week 4: number analyzed (Participants) | 76 | 77
  Work days missed at week 4 | 0.9 (1.7) | 1.2 (3.6)

ADVERSE EVENTS:
Time Frame: From time of assignment until study completion (at week 4).
Arm/Group | Intervention Arm | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT02899065/Prot_SAP_000.pdf